CLINICAL TRIAL: NCT03406416
Title: Evaluation of a Suprachoroidal Retinal Prosthesis: A 44 Channel Fully Implantable Study
Brief Title: Study of a Suprachoroidal Retinal Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mobius Medical Pty Ltd. (Industry)
Collaborators: Bionic Vision Technologies (Unknown); Center for Eye Research Australia (Other); The Bionics Institute of Australia (Other); University of Melbourne (Other); Data 61 CSIRO (Unknown); Australian National University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVT_001
Record Dates: First submitted 2017-12-26; First posted 2018-01-23 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Retinitis Pigmentosa; Choroideremia
MeSH Terms: conditions — Retinitis Pigmentosa; Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suprachoroidal retinal prosthesis (Experimental): Prototype wide view suprachoroidal retinal prosthesis
  Interventions: Device: 44Ch Bionic Eye Device

INTERVENTIONS:
Device: 44Ch Bionic Eye Device — Prototype wide view suprachoroidal retinal prosthesis

SUMMARY:
This study is a proof of principal, to evaluate a safety and efficacy of a prototype suprachoroidal retinal implant.

DETAILED DESCRIPTION:
Retinal visual prostheses are currently in early development as an intervention to improve functional vision in people who have become blind from retinal degenerative eye disease. This study follows on from an initial proof of concept study (n=3) between 2012 and 2014, and will test a second-generation retinal prosthesis device, which has the ability to be used outside of the laboratory environment (i.e. is fully implantable).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Either gender
* A confirmed history of outer retinal degenerative disease such as retinitis pigmentosa or choroideremia
* Remaining visual acuity of bare light perception or less in both eyes
* Functional inner retina (ganglion cells and optic nerve), as shown by the ability to perceive light and/or a measurable corneal electrically evoked visual response
* A history of at least 10 years of useful form vision in the worse seeing eye

Exclusion Criteria:

* Optic nerve disease (history of glaucoma of More than 1 month, or history of any other optic neuropathy)
* Diseases of the inner retina including, but not limited to, central retinal artery or vein occlusion (CRAO, CRVO), end stage diabetic retinopathy, retinal detachment, traumatic retinal damage, infectious retinal disease, inflammatory retinal disease.
* Inability to visualise the retina due to corneal or other ocular media opacities (corneal degenerations, dense cataracts, trauma, lid malpositions)
* Any ocular condition that predisposes the participant to rubbing their eyes
* Cognitive deficiencies, including dementia or progressive neurological disease
* Psychiatric disorders, including depression, as diagnosed by a qualified psychologist
* Deafness or significant hearing loss
* Inability to speak or understand English
* Pregnancy
* Presence of a cochlear implant
* Participant enrolled in another investigational drug or device trial for the treatment of their ocular condition
* Poor general health, which would exclude them from obtaining a general anaesthetic
* Unrealistic expectations of the investigational device to provide functional vision
* Poorly controlled diabetes
* Epilepsy
* Unsuitable level of regular nystagmus (which would prevent ocular images from being obtained)
* Anyone with medical devices (implanted or carried) that could cause serious health problems if compromised by electro-magnetic interference

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Number and severity of device related serious adverse events (SAEs) | 2 years
  The safety of the surgical implantation assessed by the number and severity of serious adverse events (SAEs) compared to other retinal prosthesis.

SECONDARY OUTCOMES:
Efficacy - visual response | 2 years
  The ability to generate a visual response accessed via repeatable threshold measurements of visual perception.
Visual Function and Functional Vision | 2 years
  Visual function and Functional Vision will be scored from performance on a range of acuity, orientation and mobility, and activities of daily living tasks. Outcome measures include:
  1. Grating visual acuity: record the grating acuity level and average response time.
  2. Square localization: response error and response time is measured.
  3. Motion detection: response error and response time is measured.
  4. Table top task: locate and identify objects on a table. Accuracy rates and response times will be recorded.
  5. Doorway detection task: to find doorway target. Task time and accuracy of door touch will be recorded.
  6. Obstacle avoidance task: task time and number of collisions is recorded.
  7. Functional Low Vision Observer Rated Assessment (FLORA): this assessment tool Is used to evaluate participant functional vision and mobility.
Quality of life - IVI - very low vision validated questionnaire | 2 years
  Quality of life will be assessed via survey and self-report. The Functional Low Vision Observer Assessment (FLORA) is a questionnaire that will be used to measure participants changes in participant daily living experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Penelope Allen, FRACO, FRACS, Principal Investigator — Center for Eye Research Australia
Locations (1):
- Centre for Eye Research Australia, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayton LN, Blamey PJ, Guymer RH, Luu CD, Nayagam DA, Sinclair NC, Shivdasani MN, Yeoh J, McCombe MF, Briggs RJ, Opie NL, Villalobos J, Dimitrov PN, Varsamidis M, Petoe MA, McCarthy CD, Walker JG, Barnes N, Burkitt AN, Williams CE, Shepherd RK, Allen PJ; Bionic Vision Australia Research Consortium. First-in-human trial of a novel suprachoroidal retinal prosthesis. PLoS One. 2014 Dec 18;9(12):e115239. doi: 10.1371/journal.pone.0115239. eCollection 2014. PMID 25521292
- [Derived] Abbott CJ, Baglin EK, Kolic M, McGuinness MB, Titchener SA, Young KA, Yeoh J, Luu CD, Ayton LN, Petoe MA, Allen PJ. Interobserver Agreement of Electrode to Retina Distance Measurements in a Second-Generation (44-Channel) Suprachoroidal Retinal Prosthesis. Transl Vis Sci Technol. 2022 Sep 1;11(9):4. doi: 10.1167/tvst.11.9.4. PMID 36066322
- [Derived] Titchener SA, Nayagam DAX, Kvansakul J, Kolic M, Baglin EK, Abbott CJ, McGuinness MB, Ayton LN, Luu CD, Greenstein S, Kentler WG, Shivdasani MN, Allen PJ, Petoe MA. A Second-Generation (44-Channel) Suprachoroidal Retinal Prosthesis: Long-Term Observation of the Electrode-Tissue Interface. Transl Vis Sci Technol. 2022 Jun 1;11(6):12. doi: 10.1167/tvst.11.6.12. PMID 35696133
- [Derived] Petoe MA, Titchener SA, Kolic M, Kentler WG, Abbott CJ, Nayagam DAX, Baglin EK, Kvansakul J, Barnes N, Walker JG, Epp SB, Young KA, Ayton LN, Luu CD, Allen PJ; Bionics Institute and Centre for Eye Research Australia Retinal Prosthesis Consortium. A Second-Generation (44-Channel) Suprachoroidal Retinal Prosthesis: Interim Clinical Trial Results. Transl Vis Sci Technol. 2021 Aug 12;10(10):12. doi: 10.1167/tvst.10.10.12. PMID 34581770
- [Derived] Karapanos L, Abbott CJ, Ayton LN, Kolic M, McGuinness MB, Baglin EK, Titchener SA, Kvansakul J, Johnson D, Kentler WG, Barnes N, Nayagam DAX, Allen PJ, Petoe MA. Functional Vision in the Real-World Environment With a Second-Generation (44-Channel) Suprachoroidal Retinal Prosthesis. Transl Vis Sci Technol. 2021 Aug 12;10(10):7. doi: 10.1167/tvst.10.10.7. PMID 34383875